CLINICAL TRIAL: NCT07059468
Title: Relationship Between Bilateral Femoral Neck Bone Mineral Density and Clinical Parameters in Stroke Patients
Brief Title: Osteoporosis After Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tuğba Atan, MD, Assoc. Prof, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: E-34225015 06/001; Gaziler (Other: Gaziler Fizik Tedavi ve Rehabilitasyon SUAM)
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Osteoporosis
Keywords: Stroke Osteoporosis
MeSH Terms: conditions — Stroke; Osteoporosis | interventions — Bone Density

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bone mineral density/ Bone mineral density (BMD) will be measured on the lumbar spine (L1-L4) and femoral neck by dual X-ray absorptiometry (DXA) — Bone mineral density/ Bone mineral density (BMD) will be measured on the lumbar spine (L1-L4) and femoral neck by dual X-ray absorptiometry (DXA) method

SUMMARY:
The aim of this study was to investigate the clinical features affecting bone mineral density in plegic and non-plegic extremities in hemiplegic patients with stroke in the subacute and chronic phases.

DETAILED DESCRIPTION:
One of the common complications after stroke is secondary osteoporosis that develops due to stroke. The most important event that draws attention to bone health in stroke patients is fractures, the most serious of which in terms of morbidity and mortality are hip fractures. The risk of hip fracture in stroke patients is 2-4 times higher than the normal population due to the decrease in bone mineral density on the plegic side and the increased risk of falling. There is a loss of bone mineral density after stroke. This loss is faster and larger in the early stages of stroke and is greater on the plegic side. The factors affecting this loss of bone mineral density after stroke have not been well defined. The relationship between stroke-related bone mineral density loss and motor function, functional mobility, balance, and muscle mass is not clear. It is important to reveal the changes in bone structure after stroke and the factors affecting this change. The aim of this study was to investigate the clinical features affecting bone mineral density in plegic and non-plegic extremities in hemiplegic patients with stroke in the subacute and chronic phases.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-65 years with a unilateral stroke confirmed by magnetic resonance imaging (MRI) or computed tomography (CT)
* Patients with a cognitive status sufficient to understand the study instructions (Mini-Mental State Assessment score ≥ 23)
* Patients with stable medical and psychological status
* Patients willing to participate in the study

Exclusion Criteria:

* Presence of hip pathologies that may lead to incorrect measurements in bone mineral density (advanced osteophytic coxarthrosis, heterotrophic ossification, internal fixator, etc.)
* Previous hip, lumbar vertebra fractures (osteoporotic compression fractures)
* History of multiple strokes
* History of concomitant neurological diseases other than stroke (Parkinson, multiple sclerosis, myopathy, etc.)
* History of diseases that may cause secondary osteoporosis (hypogonadism, primary hyperparathyroidism, thyrotoxicosis, malabsorption, etc.)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 44 Patients aged 40-65 years with a unilateral stroke confirmed by magnetic resonance imaging (MRI) or computed tomography (CT)
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Dual X-ray absorptiometry (DXA) | baseline
  Bone mineral density/ Bone mineral density (BMD) will be measured on the lumbar spine (L1-L4) and femoral neck by dual X-ray absorptiometry (DXA) method./ Baseline

SECONDARY OUTCOMES:
Manual muscle strength measurement/ Muscle strength | baseline
  Manual muscle strength measurement/ Muscle strength will be evaluated by the Medical Research Council muscle strength scale. This scale is a 6-point scale. (0 = no movement; 1 = tremor of movement; 2 = movement with gravity eliminated; 3 = movement against gravity; 4 = movement against resistance; 5 = full strength
Fugl-Meyer Lower Extremity Motor Subscale | baseline
  This scale evaluates motor function, sensory function, balance, range of motion, and joint pain, and the maximum score is 226. The maximum possible scores on the motor scale are 100 points for the upper (66) and lower (34) extremities, 24 for the sensory scale, 14 for balance, 44 for range of motion, and 44 for joint pain. The motor scale evaluates the mobility of the shoulder, elbow, forearm, wrist, hand, hip, knee, and ankle. Accordingly, 0 indicates that the movement cannot be performed, 1 indicates that it can be performed partially, and 2 indicates that the movement can be performed fully. The motor scale also includes reflex and coordination-speed evaluations (Gladstone et al., 2002). The motor-coordination subscale has a maximum score of 66 points for the upper extremity and a maximum score of 34 points for the lower extremity. Higher scores indicate better motor recovery. In this study, lower extremity motor subscale will be used
Functional Ambulation Classification | baseline
  The Functional Ambulation Classification is a functional walking test that evaluates ambulation ability. It includes six different categories and assesses ambulation status by determining how much support the patient needs while walking, regardless of whether they use assistive devices.
Spasticity assessment/ Ashworth graded spasticity from 0 to 4 | baseline
  . Accordingly, 0 indicates normal muscle tone, 1 indicates a slight increase in muscle tone - a feeling of catching, 2 indicates a more pronounced increase in muscle tone (the extremity can be easily moved), 3 indicates a marked increase in muscle tone, and 4 indicates a rigid joint.
Berg Balance Scale | baseline
  The Berg Balance Scale is a widely used clinical test that can reveal a person's static and dynamic balance abilities. Total test score range from 0 (lowest balance) to 56 (highest balance) ability.
International Fall Activity Scale | baseline
  The International Fall Activity Scale is a scale that examines an individual's concerns about the possibility of falling during 16 different activities that do not threaten daily life.The response option ranged from 1-4 depicted by 1 for being not at all concerned, 2 for being somewhat concerned, 3 for being fairly concerned and 4 for being very concerned.
Ultrasonographic evaluation | baseline
  Ultrasonographic evaluation of quadriceps femoris muscle thickness

CONTACTS AND LOCATIONS:
Overall Officials: Engin Koyuncu, Prof., Study Director — SBÜ ANKARA GAZİLER FİZİK TEDAVİ VE REHABİLİTASYON EĞİTİM VE ARAŞTIRMA HASTANESİ
Locations (1):
- Sbü Ankara Gaziler Fizik Tedavi Ve Rehabilitasyon Eğitim Ve Araştirma Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No